CLINICAL TRIAL: NCT07174037
Title: Impact of Planter Flexors Spasticity on Postrual Stabilty and Functional Outcome in Pateints With Stroke
Acronym: PFS
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Shokry Abd Elmotaleb Ameen, principle investigator : radwa shokry abd-elmotaleb ameen, Cairo University
Other Study IDs: P.T.REC/012/005968
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Planter Flexors Spasticity; Postrual Stabilty; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low spasticity group: thirty four patients with low spasticity grade (grade I and 2) will participate in this group
  Interventions: Other: Low spasticity group
- High spasticity group: thirty four patients with high spasticity grade (grade 3 and 4) will participate in this group
  Interventions: Other: High spasticity group

INTERVENTIONS:
Other: Low spasticity group — low sapsticity (grade 1-2) unilateral ischemic stroke will be participate in this group
  Groups: Low spasticity group
Other: High spasticity group — high sapsticity (grade 3-4) unilateral ischemic stroke will be participate in this group
  Groups: High spasticity group

SUMMARY:
this study will be conducted to investigate the effect of planter flexors spasticity on postural stability, risk of falling and function outcomes in patients with stroke

DETAILED DESCRIPTION:
Lower limb spasticity is a common following a cerebrovascular attack (CVA) or stroke, which can affect the balance and gait of patients. This then not only affects independence, and quality of life but increases the risk for other concerns, such as falling and an increased sedentariness, which could further affect health outcomes.The spasticity of the planter flexors disturbs walking, can impede toe clearance during the swing phase of gait causing the patient to fall as a result their toe 'catching' on the ground .In stroke patients characteristically the extensors of the leg are spastic and the flexors are weak . All these changes lead to gait disturbance as well as impaired functional mobility of patients.Studies have shown that patients with stroke have a higher risk of developing the fear of falling, which may be related to an increased risk of falling after stroke .The incidence of fear of falling after stroke has been reported to be approximately 32 to 66 percent. Fear of falling is associated with adverse consequences such as limited activity, increased incidence of falls, decreased quality of life, and increased hospitalization and case fatality rates

ELIGIBILITY:
Inclusion Criteria:

* Sixty eight first-ever unilateral ischemic stroke patients as diagnosed by CT ''computed topography'' or MRI ''magnetic resonance imaging.
* Patients will be both sexes.
* Their age ranges from 45 to 60 years
* The patients will be divided into 2 groups based on their level of ankle plantar flexor spasticity according to the Modified Ashworth Scale (MAS):
* Low spasticity (grade 1 and 1+).
* High spasticity (grade 2 and 3).
* Duration of illness will be over 6 months post-stroke.
* Body mass index of patients will be ≤ 30 kg / m2
* Patients can stand independently.
* Normal cognitive abilities according to MOKA scale will be ≥ 24

Exclusion Criteria:

* Bilateral hemiplegia.
* Patients having any other neurological disorders affecting their lower limb extremity as MS, Parkinson disease, peripheral neuropathy.
* Patients with visual auditory impairment affecting their ability to complete task. 4.Patients with previous fracture of the lower limbs or any other musculoskeletal disorders such as severe arthritis, fixed ankle contracture, ankle surgery, leg length discrepancy or being treated with botulinum toxin injections within the past 3 months of study participation.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sixty eight unilateral ischemic stroke patients as diagnosed by CT ''computed topography'' or MRI ''magnetic resonance imaging from both sexes and will be assigned to two groups depending on level of spasticity.
  * Low spasticity (grade 1 and 1+).
  * High spasticity (grade 2 and 3).
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
spasticity | up to thirty minutes
  Modified Ashworth scale will be used to assess spasticity.The rater will score muscle spasticity from 0 to 4. Only one passive stretch will be applied to rate spasticity
  The scale is as follows:
  0: No increase in muscle tone
  1. Slight increase in muscle tone, with a catch and release or minimal resistance at the end of the range of motion when an affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested as a catch, followed by minimal resistance through the remainder (less than half) of the range of motion
  2. A marked increase in muscle tone throughout most of the range of motion, but affected part(s) are still easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
muscle spasticity | up to thirty minutes
  MyotonPRO will be used to assess spasticity. it can assess regional differences in tendon stiffness, such as variations along the Achilles tendon, and monitor stiffness modulation with joint position changes.
  It is placed on the skin over the muscle. A brief, gentle tap from the probe causes the muscle to oscillate. The oscillations are analysed automatically by the device to calculate the muscle's mechanical characteristics, such as its tone, stiffness and how elastic it is.
postural stability | up to thirty minutes
  biodex balance system will be used to assess postural stability
risk of falling index | up to thirty minutes
  biodex balance system will be used to assess risk of falling
risk of falling | up to thirty minutes
  The Morse Fall Scale (MFS) is one of the well- known tools both domestically and internationally for measuring fall risk in adults. It has the advantage of being easy to measure. The MFS has been validated in several studies and is considered a reliable tool for measuring fall risk. The MFS is composed of six variables that assess different risk factors for falling. Each variable is scored, and the total score determines the patient's fall risk.Each of the six variables is assigned a score, and the total score ranges from 0 to 125. The risk levels are categorized as follows:
  Low Risk: 0-24 Moderate Risk: 25-44 High Risk: 45 and above
functional mobility | up to thirty minutes
  The Timed Up and Go (TUG) test is a widely utilized clinical tool to assess functional Mobility.It involves timing an individual as they stand up from a chair with armrests, walk a distance of three meters at a comfortable place (with or without their usual walking aid), turn around, walk back, and sit down again
  * 10 seconds: Normal mobility.
  * 20 seconds: Good mobility, able to go out alone without gait aid.
  * 30 seconds: Mobility problems, requires gait aid, cannot go outside alone.
    * 14 seconds indicates a high risk of falls.